CLINICAL TRIAL: NCT07114757
Title: REnal Denervation After Stroke (REDs) Study - A Randomized Clinical Trial of Renal Denervation in the Subacute Phase of Stroke
Acronym: REDs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro per la Lotta Contro l'Infarto - Fondazione Onlus (Other)
Responsible Party: Principal Investigator, Francesco Versaci, Chief of Cardiology, Ospedale Santa Maria Goretti
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDs
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Disease; Arterial Hypertension; Hypertension; Renal Denervation; Stroke
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders; Hypertension; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RDN (Experimental): This arm includes the patients who will be treated with renal denervation.
  Interventions: Procedure: Renal denervation after stroke
- Standard therapy (No Intervention): This arm includes the patients who will be treated with standard therapy.

INTERVENTIONS:
Procedure: Renal denervation after stroke — Renal sympathetic denervation (RDN) is a minimally invasive catheter-based procedure targeting renal sympathetic nerve fibers to achieve sustained reductions in blood pressure.
  Arms: RDN

SUMMARY:
The REnal Denervation after stroke (REDs) study is a national, multicenter, investigator-initiated randomized controlled clinical trial designed to assess the efficacy of catheter-based renal denervation (RDN) performed in the subacute phase of stroke among patients with drug-resistant hypertension. Conducted across 15 Italian centers, this pragmatic trial adopts a parallel-group design with participants randomized in a 1:1 ratio to receive either RDN using the Symplicity Spyral system or standard care. Randomization will occur via a secure online platform, and the intervention will be performed within 24 hours post-randomization, adhering to a standardized procedural protocol.

The trial targets adult patients aged 18 to 84 years who have experienced a stroke 7 to 45 days prior to enrollment and present with persistent systolic hypertension (≥140 mmHg) or a non-dipping profile on ambulatory blood pressure monitoring, despite the use of at least two antihypertensive medications at maximum tolerated doses. Following informed consent and verification of eligibility, enrolled patients will undergo baseline assessments including physical examination, laboratory testing, ECG, stroke severity and disability scoring, and quality of life evaluation.

The total duration of the REDs study is 48 months, encompassing a 24-month enrollment window and a 24-month follow-up period. Study endpoints, including 24-hour ambulatory blood pressure and secondary clinical and functional outcomes, will be evaluated at 3, 6, 9, 12, and 24 months following the intervention. These follow-up assessments will be conducted through hospital visits or teleconsultations as appropriate.

The primary efficacy endpoint is the change in mean 24-hour systolic blood pressure 12 months after randomization. Secondary endpoints include diastolic and mean arterial pressure, antihypertensive medication burden, time to blood pressure control, functional neurological scores (NIHSS, mRS), quality of life metrics, and stroke recurrence. Data collection will be managed via an electronic case report form (eCRF), and adverse events will be monitored throughout the study in line with ISO14155 and GCP standards.

This trial is supported by an unrestricted grant from Medtronic and adheres to ethical guidelines as outlined by the Declaration of Helsinki and GDPR. The REDs study aims to generate clinically relevant evidence to support the integration of RDN into secondary prevention strategies for stroke patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

- We will enroll patients (at least 18 years of age and younger than 85 years old) with subacute stroke (thus occurring 7-45 days before screening), admitted to hospital, with persistently high systolic PB (≥140 mm Hg computed as the mean of 3 repeated measurements taken within 5 minutes between 8.00am and 8.30 am on 2 consecutive days, thus totaling 6 measurements), or a non-dipper profile at ambulatory BP monitoring, despite therapy with ≥2 anti-hypertensive drugs at maximum tolerated dose. Patients should be medically stable with no severe complications such as infections, or worsening of neurological status that would require immediate and intensive medical or surgical intervention.

Exclusion Criteria:

* ⦁ Patients with cerebral bleeding due to arteriovenous malformation or intracranial aneurysm

  * Hemodynamic instability
  * Comorbidity with life expectancy ≤ 1 year
  * Renal artery anatomy, which prevents the procedure
  * Reno vascular disease
  * Vascular occlusion, which prevents the procedure
  * Secondary hypertension
  * Subject has known hypersensitivity or contraindication to any of the study drugs
  * The subject is currently participating in another investigational drug or device clinical study
  * Pregnancy or nursing
  * Presence of other anatomic or comorbid conditions or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements or impact the scientific soundness of the clinical investigation results

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2027-09-25 (Estimated); Study Completion 2029-09-25 (Estimated)

PRIMARY OUTCOMES:
mean 24-hour systolic blood pressure 12 months after randomization | 12 months
  mean 24-hour systolic blood pressure 12 months after randomization

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Maria Goretti Hospital, Latina, LT, Italy